CLINICAL TRIAL: NCT06091943
Title: Phase 1 Study to Evaluate the Bioavailability of Tislelizumab Via Subcutaneous Injection in the First-Line Treatment of Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study to Evaluate the Bioavailability of Tislelizumab Via Subcutaneous Injection in First-Line Treatment of Participants With Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-103; CTR20233814 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose/Injection Site Exploration (Experimental): Different injection sites will be evaluated; participants will receive tislelizumab in predefined administration sequences plus histology-based chemotherapy consisting of either cisplatin/carboplatin and pemetrexed or carboplatin and paclitaxel/nab-paclitaxel depending on the cancer subtype.
  Interventions: Drug: Tislelizumab IV; Drug: Tislelizumab SC; Drug: Histology-Based Chemotherapy Doublet
- Part 2: Dose Expansion (Experimental): The recommended dose of tislelizumab SC determined from Part 1 plus histology-based chemotherapy consisting of either cisplatin/carboplatin and pemetrexed or carboplatin and paclitaxel/nab-paclitaxel depending on the cancer subtype will be evaluated.
  Interventions: Drug: Tislelizumab SC; Drug: Histology-Based Chemotherapy Doublet

INTERVENTIONS:
Drug: Tislelizumab IV — Planned doses will be administered intravenously.
  Other Names: BGB-A317 IV
  Arms: Part 1: Dose/Injection Site Exploration
Drug: Tislelizumab SC — Planned doses will be administered via subcutaneous injection.
  Other Names: BGB-A317 SC
Drug: Histology-Based Chemotherapy Doublet — Chemotherapy Doublet 1: Cisplatin/carboplatin + pemetrexed.
  Chemotherapy Doublet 2: Carboplatin + paclitaxel/nab-paclitaxel.
  Choice of histology-based induction chemotherapy doublet will be determined by the investigator and will be administered at standard doses intravenously.

SUMMARY:
This is an open-label, multicenter, Phase 1 clinical study to evaluate the bioavailability of tislelizumab subcutaneous (SC) injection in the first-line treatment of participants with advanced or metastatic non-small cell lung cancer (NSCLC). This clinical study will be divided into 2 parts: dose/injection site exploration (Part 1) and dose expansion (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Able to sign a written consent form, understand, and agree to comply with requirements of the study.
* Documented locally advanced or recurrent NSCLC that is not eligible for curative surgery and/or definitive radiotherapy, with or without chemotherapy, or metastatic non-squamous or squamous NSCLC.
* No prior systemic treatment for advanced or metastatic NSCLC, including but not limited to chemotherapy or targeted therapy.
* At least one measurable lesion as assessed by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) PS ≤ 1.
* Adequate organ function as indicated by laboratory tests.

Exclusion Criteria:

* Participants diagnosed with NSCLC that harbor a driver mutation (eg, EGFR-sensitizing mutation, ALK fusion oncogene, and BRAF V600E mutation or ROS1 mutation).
* Participant has received any Chinese herbal medicine or Chinese patent medicines used to control cancer within 14 days before first dose of study drug.
* Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
* Active autoimmune diseases or history of autoimmune diseases that may relapse.
* Any cancer ≤ 5 years before first dose of study drug except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, localized prostate cancer, carcinoma in situ of the cervix or breast).
* Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before first dose of study drug.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Area under the concentration-time curve (AUC) of Tislelizumab SC | Up to approximately 3.5 months
Part 1 and 2: Concentration at the end of dosing interval (Ctrough) of Tislelizumab SC | Up to approximately 3.5 months
Part 1: Bioavailability of Tislelizumab SC | Up to approximately 2 months
Part 2: Maximum observed plasma concentration (Cmax) of Tislelizumab SC | Up to approximately 3.5 months
Part 2: Accumulation ratio (Rac) of Tislelizumab SC | Up to approximately 3.5 months
Part 2: Elimination half-life (t1/2) of Tislelizumab SC | Up to approximately 3.5 months
Part 2: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 27 months
  Number of participants with AEs and SAEs and laboratory abnormalities, reported during the AE reporting period and characterized by type, frequency, severity (as graded by National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0 [NCI-CTCAE v5.0]), timing, seriousness, and relationship to study therapy.

SECONDARY OUTCOMES:
Part 1: Maximum observed concentration (Cmax) of Tislelizumab SC | Up to approximately 2 months
Part 1: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 27 months
  Number of participants with AEs and SAEs and laboratory abnormalities, reported during the AE reporting period and characterized by type, frequency, severity (as graded by NCI-CTCAE v5.0), timing, seriousness, and relationship to study therapy.
Part 1 and 2: Number of Participants with Anti-Tislelizumab Antibodies | Up to 25 months
Part 2: Overall Response Rate (ORR) of Tislelizumab SC | Up to approximately 27 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as determined from tumor assessments by investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1).
Part 2: Duration of Response (DOR) of Tislelizumab SC | Up to approximately 27 months
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death due to any cause, whichever occurs first as assessed by the investigator.
Part 2: Progression-Free Survival (PFS) | Up to approximately 27 months
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (15):
- China (13):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Jining No Peoples Hospital East Branch, Jining, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Deyangs People Hospital, Deyang, Sichuan
  - Huzhou Central Hospital, Huzhou, Zhejiang
- Arensia Exploratory Medicine Llc, Tbilisi, Georgia
- The Institute of Oncology, Arensia Exploratory Medicine, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/